CLINICAL TRIAL: NCT00826540
Title: Phase II Study of Sorafenib/Avastin® as Salvage Therapy in Patients With Metastatic Colorectal Cancer
Brief Title: Sorafenib and Bevacizumab in Treating Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N054C; NCI-2009-01177 (Registry Identifier: CTRP (Clinical Trials Reporting System)); U10CA025224 (NIH); CDR0000632342 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2009-01-21; First posted 2009-01-22 (Estimated); Results first posted 2014-03-03 (Estimated); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Recurrent Colon Cancer; Recurrent Rectal Cancer; Stage IV Colon Cancer; Stage IV Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Sorafenib; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (sorafenib tosylate and bevacizumab) (Experimental): Patients receive sorafenib tosylate orally twice daily on days 1-5 and 8-12 and bevacizumab IV over 30-90 minutes on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity. Blood samples are collected at baseline and then periodically during study treatment for laboratory biomarker and pharmacogenetic studies
  Interventions: Drug: sorafenib tosylate; Biological: bevacizumab

INTERVENTIONS:
Drug: sorafenib tosylate — Given orally
  Other Names: BAY 43-9006; BAY 43-9006 Tosylate Salt; BAY 54-9085; Nexavar; SFN
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF

SUMMARY:
This phase II trial is studying how well giving sorafenib together with bevacizumab works in treating patients with metastatic colorectal cancer. Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Sorafenib and bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Giving sorafenib together with bevacizumab may kill more tumor cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate proportion of patients who are progression-free at 3 months (in historic comparison with results for single-agent bevacizumab in ECOG 3200).

SECONDARY OBJECTIVES:

I. Response rate (RR) II. Overall survival (OS) III. Safety IV. Feasibility

OUTLINE: This is a multicenter study.

Patients receive sorafenib tosylate orally twice daily on days 1-5 and 8-12 and bevacizumab IV over 30-90 minutes on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity. Blood samples are collected at baseline and then periodically during study treatment for laboratory biomarker and pharmacogenetic studies.

After completion of study treatment, patients are followed periodically for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stage IV colorectal cancer (histologic proof is not required)
* Measurable disease

  * Spiral CT scan required for both pre- and post-treatment tumor assessments of lesions measuring 1-2 cm
* Progressive disease during or within 6 months of most recent prior chemotherapy regimen (bevacizumab, fluoropyrimidine, oxaliplatin, or irinotecan-based treatment) OR considered ineligible for standard therapy
* Documentation of submission of tumor material for Kirsten Rat Sarcoma (KRAS) testing available
* Prior anti-epidermal growth factor receptor (EGFR) antibody therapy (e.g., cetuximab or panitumumab) required for patients with wild-type KRAS tumor
* No known brain metastasis

  * Patients with neurological symptoms must undergo a CT scan or MRI of the brain to exclude brain metastasis
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Life expectancy ≥ 6 months
* Hemoglobin ≥ 9.0 g/dL
* Absolute neutrophil count (ANC) ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* White blood cell count (WBC) ≥ 3,400/mm³
* International normalized ratio (INR) < 1.5 (≤ 3.0 if on anti-coagulation therapy [e.g., warfarin or heparin])
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Aspartate aminotransferase (AST) ≤ 2.5 times ULN (≤ 5 times ULN if there is liver involvement)
* Alkaline phosphatase ≤ 3 times ULN
* Creatinine ≤ 1.5 times ULN
* Urine protein:creatinine ratio < 1 OR urine dipstick < 2+ OR urine protein < 1,000 mg by 24-hour urine collection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 6 months after completion of study treatment (≥ 2 weeks after completion of treatment with sorafenib tosylate alone)
* Willing to provide mandatory blood samples for translational research studies
* Able to swallow whole pills
* No inadequately controlled hypertension (i.e., systolic BP > 150 mm Hg or diastolic BP > 100 mm Hg on anti-hypertensive medications)
* No prior hypertensive crisis or hypertensive encephalopathy
* No myocardial infarction or unstable angina within the past 6 months
* No congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* No thrombolic or embolic events (e.g., cerebrovascular accident, including transient ischemic attacks) within the past 6 months
* No hemorrhage or bleeding event > grade 3 within the past 4 weeks
* No evidence or history of bleeding diathesis or coagulopathy (in the absence of therapeutic anticoagulation)
* No greater than normal risk of bleeding
* No active or recent hemoptysis (≥ ½ teaspoon of bright red blood per episode) within the past 30 days
* No concurrent uncontrolled illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia requiring anti-arrhythmic drugs
  * Psychiatric illness or social situations that would limit compliance with study requirements
* No known HIV infection or chronic hepatitis B or C infection
* No serious, non-healing wound, active ulcer, or untreated bone fracture

  * Patients with fractures secondary to metastatic disease are eligible after appropriate radiotherapy
* No significant traumatic injury within the past 4 weeks
* No known or suspected allergy or hypersensitivity to any component of bevacizumab, sorafenib tosylate, or their excipients or to any other agent given in the course of this study
* No malabsorption problem
* None of the following within the past 6 months:

  * Significant vascular disease (e.g., aortic aneurysm or aortic dissection)
  * Peripheral arterial thrombosis
  * Symptomatic peripheral vascular disease
  * Abdominal fistula
  * Gastrointestinal perforation
  * Intra-abdominal abscess
* No other active malignancy within the past 3 years except non melanoma skin cancer or carcinoma in situ of the cervix

  * Prior malignancy allowed provided patient is not receiving other specific treatment for that malignancy (other than hormonal therapy)
* No other concurrent investigational agent for this cancer
* Prior radiotherapy allowed
* No prior sorafenib tosylate
* No prior discontinuation of bevacizumab due to adverse events
* More than 4 weeks since prior and no concurrent participation in any other experimental drug study
* More than 4 weeks since prior St. John's wort or rifampin
* More than 4 weeks since prior and no concurrent major surgical procedure or open biopsy
* More than 7 days since prior core biopsy or minor surgical procedure, including placement of a vascular access device
* No concurrent anticoagulant, except low-dose warfarin or heparin for deep venous thrombosis prophylaxis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2010-01 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Axel Grothey, MD, Study Chair — North Central Cancer Treatment Group
Locations (211):
- United States (211):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Saint Anthony Central Hospital, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Exempla Saint Joseph Hospital, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program CCOP, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Galesburg Clinic, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael MD (UIA Investigator), Moline, Illinois
  - Sharis, Christine M MD (UIA Investigator), Moline, Illinois
  - Stoffel, Thomas J MD (UIA Investigator), Moline, Illinois
  - Holy Family Medical Center, Monmouth, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Pekin Cancer Treatment Center, Pekin, Illinois
  - Pekin Hospital, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois Oncology Research Association CCOP, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Saint Margaret's Hospital, Spring Valley, Illinois
  - Saint Francis Hospital and Health Centers, Beech Grove, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - Indiana University Health La Porte Hospital, La Porte, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Reid Hospital and Health Care Services, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - Cedar Rapids Oncology Association, Cedar Rapids, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Capitol, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa Oncology Research Association CCOP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Siouxland Hematology Oncology Associates, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Hospital District Sixth of Harper County, Anthony, Kansas
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Main Office, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita CCOP, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium Community Clinical Oncology Program, Ann Arbor, Michigan
  - Oakwood Hospital, Dearborn, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Allegiance Health, Jackson, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Lakeland Hospital, Saint Joseph, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Sanford Clinic North-Bemidgi, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Duluth Clinic CCOP, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Immanuel-Saint Joseph Hospital-Mayo Health System, Mankato, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Metro-Minnesota CCOP, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology and Hematology PA-Woodbury, Woodbury, Minnesota
  - Saint John's Hospital, Springfield, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Center for Cancer Care and Research, St Louis, Missouri
  - Montana Cancer Consortium CCOP, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies PC, Billings, Montana
  - Billings Clinic, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Hospital, Missoula, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Sanford Medical Center-Fargo, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - North Coast Cancer Care-Clyde, Clyde, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Dayton CCOP, Dayton, Ohio
  - Hematology Oncology Center Incorporated, Elyria, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Saint Luke's Hospital, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Cancer Center at Saint Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Adventist Medical Center, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazelton, Hazleton, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley, Wilkes-Barre, Pennsylvania
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Midelfort Clinic-Clairemont Campus, Eau Claire, Wisconsin
  - Mayo Clinic Health System Eau Claire Hospital - Luther Campus, Eau Claire, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Mary's Hospital, Green Bay, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Green Bay Oncology - Oconto Falls, Oconto Falls, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Derived] Xie H, Lafky JM, Morlan BW, Stella PJ, Dakhil SR, Gross GG, Loui WS, Hubbard JM, Alberts SR, Grothey A. Dual VEGF inhibition with sorafenib and bevacizumab as salvage therapy in metastatic colorectal cancer: results of the phase II North Central Cancer Treatment Group study N054C (Alliance). Ther Adv Med Oncol. 2020 Mar 6;12:1758835920910913. doi: 10.1177/1758835920910913. eCollection 2020. PMID 32201506

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 83 patients were registered between 06/03/2009 and 10/20/2009 from 25 North Central Cancer Treatment Group (NCCTG) sites.
Pre-assignment Details: One patient withdrew from the study and three patients were ineligible, therefore, these patients were excluded from all results.
Groups:
- Treatment (Sorafenib Tosylate and Bevacizumab): Patients receive sorafenib tosylate orally twice daily on days 1-5 and 8-12 and bevacizumab IV over 30-90 minutes on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity. Blood samples are collected at baseline and then periodically during study treatment for laboratory biomarker and pharmacogenetic studies> > sorafenib tosylate: Given orally>
  > bevacizumab: Given IV
Period: Overall Study
Arm/Group | Treatment (Sorafenib Tosylate and Bevacizumab)
Started | 83
Completed | 79
Not Completed | 4
Not completed — ineligible | 3
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Sorafenib Tosylate and Bevacizumab)
Number analyzed (Participants) | 79
Age, Continuous [Median (Full Range); unit: years] | 62 [36 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 43
Performance Score [Number; unit: participants] — The Eastern Cooperative Oncology Group (ECOG) performance score, runs from 0 to 5, with 0 denoting perfect health and 5 death.
  participants
    0 (Fully active) | 44
    1 (Restricted in physically strenuous activity) | 35
Kirsten rat sarcoma (KRAS) [Number; unit: participants]
  Wild-type | 39
  Mutated | 40

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival Rate
Description: The primary endpoint of this trial is progression free survival at 3 months. All patients meeting the eligibility criteria who have signed a consent form and have begun treatment will be considered evaluable. Patients lost to follow-up before 3 months (e.g., progression, refusing further treatment, etc.) will be considered treatment failures. All eligible patients will be followed until death or a minimum of 3 years. The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients.
  Progression is defined as at least a 20% increase in the sum of longest liameter of target lesions taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: At 3 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Treatment (Sorafenib Tosylate and Bevacizumab): Patients receive sorafenib tosylate orally twice daily on days 1-5 and 8-12 and bevacizumab IV over 30-90 minutes on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity. Blood samples are collected at baseline and then periodically during study treatment for laboratory biomarker and pharmacogenetic studies >
  > sorafenib tosylate: Given orally
  >
  > bevacizumab: Given IV
Arm/Group | Treatment (Sorafenib Tosylate and Bevacizumab)
Number analyzed (Participants) | 79
percentage of participants | 53.2 [41.7 to 64.4]

2. Secondary Outcome: Response Rate
Description: Number of patients reporting a partial response or complete response while on treatment
Time Frame: 2 years
Population: Only patients with one or more post-baseline disease assessments were included in analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Sorafenib Tosylate and Bevacizumab)
Number analyzed (Participants) | 73
Participants | 1

3. Secondary Outcome: Overall Survival
Description: The distribution of overall survival will be estimated using Kaplan-Meier methodology.
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Sorafenib Tosylate and Bevacizumab)
Number analyzed (Participants) | 79
months | 8.3 [5.5 to 11.3]

4. Secondary Outcome: Feasibility of Study Treatment
Description: Will be evaluated based on the number of patients who delayed treatment, omitted doses of treatment, or reduced treatment dose.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Sorafenib Tosylate and Bevacizumab)
Number analyzed (Participants) | 79
Participants
  Delayed treatment at least once | 31
  Omitted a dose of BEV at least once | 13
  Omitted a dose of sorafenib at least once | 26
  Reduced sorafenib at least once | 49

ADVERSE EVENTS:
Arm/Group | Treatment (Sorafenib Tosylate and Bevacizumab)
Serious Adverse Events (participants affected / at risk) | 13/79
Other Adverse Events (participants affected / at risk) | 78/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Sorafenib Tosylate and Bevacizumab) (N=79)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Esophageal varices hemorrhage (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Rectal fistula (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Amylase increased (Investigations) | 1 (1)
Bilirubin increased (Investigations) | 1 (1)
Cardiac troponin I increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 2 (2)
Lipase increased (Investigations) | 2 (2)
Weight loss (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 3 (3)
Thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Sorafenib Tosylate and Bevacizumab) (N=79)
Hemoglobin decreased (Blood and lymphatic system disorders) | 5 (9)
Left ventricular dysfunction (Cardiac disorders) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1)
Myocardial ischemia (Cardiac disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 37 (119)
Ascites (Gastrointestinal disorders) | 1 (2)
Colitis (Gastrointestinal disorders) | 1 (1)
Colonic obstruction (Gastrointestinal disorders) | 1 (2)
Colonic perforation (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (6)
Diarrhea (Gastrointestinal disorders) | 49 (172)
Dyspepsia (Gastrointestinal disorders) | 1 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 22 (56)
Flatulence (Gastrointestinal disorders) | 2 (7)
Mucositis oral (Gastrointestinal disorders) | 23 (53)
Nausea (Gastrointestinal disorders) | 37 (100)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Small intestinal necrosis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 19 (61)
Disease progression (General disorders) | 1 (1)
Edema limbs (General disorders) | 2 (2)
Fatigue (General disorders) | 74 (355)
Fever (General disorders) | 3 (3)
General symptom (General disorders) | 1 (1)
Pain (General disorders) | 2 (6)
Abdominal infection (Infections and infestations) | 3 (4)
Urinary tract infection (Infections and infestations) | 3 (3)
Wound dehiscence (Injury, poisoning and procedural complications) | 2 (2)
Alanine aminotransferase increased (Investigations) | 3 (6)
Alkaline phosphatase increased (Investigations) | 10 (29)
Amylase increased (Investigations) | 4 (8)
Aspartate aminotransferase increased (Investigations) | 7 (22)
Bilirubin increased (Investigations) | 4 (11)
Creatinine increased (Investigations) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 1 (2)
Leukocyte count decreased (Investigations) | 1 (6)
Lipase increased (Investigations) | 7 (19)
Lymphocyte count decreased (Investigations) | 5 (8)
Neutrophil count decreased (Investigations) | 2 (6)
Platelet count decreased (Investigations) | 3 (19)
Weight loss (Investigations) | 45 (193)
Anorexia (Metabolism and nutrition disorders) | 58 (198)
Blood glucose increased (Metabolism and nutrition disorders) | 6 (14)
Dehydration (Metabolism and nutrition disorders) | 3 (4)
Serum albumin decreased (Metabolism and nutrition disorders) | 7 (20)
Serum calcium decreased (Metabolism and nutrition disorders) | 4 (12)
Serum calcium increased (Metabolism and nutrition disorders) | 1 (2)
Serum glucose decreased (Metabolism and nutrition disorders) | 1 (1)
Serum phosphate decreased (Metabolism and nutrition disorders) | 3 (4)
Serum potassium decreased (Metabolism and nutrition disorders) | 2 (2)
Serum potassium increased (Metabolism and nutrition disorders) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 4 (14)
Serum sodium increased (Metabolism and nutrition disorders) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (15)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Joint pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (4)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (8)
Taste alteration (Nervous system disorders) | 2 (4)
Glomerular filtration rate decreased (Renal and urinary disorders) | 1 (1)
Protein urine positive (Renal and urinary disorders) | 40 (132)
Renal failure (Renal and urinary disorders) | 2 (2)
Ureteric obstruction (Renal and urinary disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Scrotal pain (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal examination abnormal (Respiratory, thoracic and mediastinal disorders) | 5 (8)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 6 (10)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (3)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 38 (169)
Rash desquamating (Skin and subcutaneous tissue disorders) | 24 (71)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 43 (146)
Hypotension (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes